| ı | FO | R | Λ | Λ. | <b>-S</b> 1 | ΓΔ | T- | N | 4 | Δ | _( | N | 1 | |
|---|----|---|-----|----|-------------|----|----|---|---|---|-----|---|---|---|
| | | | · · | 40 | -J | | | v | _ | _ | \—\ | u | _ | _ |

Version 1.0

# **Statistical Analysis Plan**

# 01\_resiLIR\_HCP

A Randomized Controlled Study to Evaluate the Feasibility and Efficacy of an Online Resilience Intervention for Healthcare Professionals ("resiLIR Healthcare Professionals")

## **Document Version History**

| Version Date | Version | Author | Signature | Change Description | Reason/Comment |
|---|---|---|---|---|---|
| 17.03.2023 | 1 | Leibniz-<br>Institute for<br>Resilience<br>Research | | Initial release. | Not applicable. |

# **TABLE OF CONTENTS**

| LIST OF | - ABBREVIATIONS | 3 |
|---------|-------------------------------------|----|
| 1. | STUDY OBJECTIVES | 4 |
| 1.1. | PRIMARY OBJECTIVE | |
| 1.2. | | |
| 2. | BACKGROUND/INTRODUCTION | 4 |
| 2.1. | STUDY DESIGN | |
| 2.2. | TREATMENT GROUPS | 4 |
| 2.3. | STUDY POPULATION | |
| 2.4. | INTERVENTION | 5 |
| 2.5. | SAMPLE SIZE | 5 |
| 2.6. | STUDY PROCEDURE | |
| 3. | POPULATIONS OF ANALYSIS | 7 |
| 4. | OUTCOME VARIABLES | 7 |
| 4.1. | PRIMARY OUTCOME | 8 |
| 4.2. | SECONDARY PARAMETERS OUTCOMES | |
| 4.3. | OTHER PARAMETERS | 9 |
| 5. | STATISTICAL METHODOLOGY | 12 |
| 5.1. | GENERAL METHODOLOGY | 12 |
| 5.2 | PRIMARY AND SECONDARY DATA ANALYSES | 12 |

## **LIST OF ABBREVIATIONS**

IG Intervention group

CG/ WLC (Waitlist-) Control group

ITT Intention-to-treat

PP Per-Protocol

ANCOVA ANalysis of COVAriance
ANOVA ANalysis Of VAriance
SD Standard Deviation

SE Standard Error

## 1. STUDY OBJECTIVES

### 1.1. PRIMARY OBJECTIVE

The goal of this clinical trial is to examine the efficacy of a newly developed online resilience intervention "resiLIR Health Care Professionals" for Health Care professionals and foster resilience in the targeted population.

#### 1.2. SECONDARY OBJECTIVES

Secondary objectives are to find out whether the intervention is effective in increasing the addressed health-related and resilience factors (e.g., optimism) as well as decreasing self-evaluations of psychopathological indicators (e.g., depression, anxiety) in healthcare professionals. Also, the study investigates whether different interventions are effective in changing state-measures of health-related self-evaluations.

Another objective is to investigate these effects in the long term (up to one-year post-intervention).

Additionally, feasibility and usability of the intervention and the newly developed platform resiLIR will be investigated.

Further objectives are to examine exploratorily the influence of the intervention on other resilience-related outcomes, mental health literacy, health seeking behaviour and stigma against mental illness and to conduct network analyses.

## 2. BACKGROUND/INTRODUCTION

Acute and chronic stress in everyday life plays an essential role in the onset and development of several physical and mental health conditions. The ability to maintain or return to mental health during stress exposure is characterized as resilience. Especially the COVID-19 pandemic emphasized the role of resilience for mental health and pointed to the importance of easily accessible and flexible interventions to improve resilience for vulnerable groups such as healthcare professionals.

### 2.1. STUDY DESIGN

Randomized Controlled Trial with 240 participants working as healthcare professionals (120 in intervention, 120 in waitlist control group), monocentric study, duration: 14 months, study design chosen to evaluate long-term effects of our training)

### 2.2. TREATMENT GROUPS

Treatment: Participants in the intervention group will gain access to the 6-week online resilience intervention "resiLIR Healthcare Professionals".

The waitlist control group will receive access to the intervention after the first follow-up assessment (3 months post-intervention).

Randomisation process: Stratified randomization is used, with age and gender as influencing factors. Randomization is performed using randomized numbers generated with Microsoft Excel. Due to the nature of the intervention, no blinding and subject replacements are planned.

Subject replacement: not applicable.

### 2.3. STUDY POPULATION

#### Inclusion criteria:

- Age 18 years or older
- Fluent in German language
- Access to web-enabled devices (tablet/laptop/computer)
- Smartphone with internet access
- Trained and employed as health care professionals
  - We used the following definition of healthcare professionals: "Healthcare professionals are specifically trained, often regulated professions that advise on or provide health services. This includes, amongst others, medical doctors, nurses, physiotherapists, speech therapists, psychotherapists, dentists, medical-technical assistants, geriatric nurses,…"

#### **Exclusion Criteria:**

- Acute mental health crisis (e.g., suicidality)
- Psychiatric/psychotherapeutic treatment
- Neurodegenerative disease(s)
- Diagnosis of schizophrenia or other psychotic disorders, bipolar disorder, post-traumatic stress disorder

## 2.4. INTERVENTION

Behavioral intervention delivered via computer/laptop and smartphone

- Weeks 1 and 2 (delivered mainly via computer): Theoretical part on stress, resilience, selfcare, and self-compassion
- Weeks 3 to 6 (delivered mainly via smartphone): Training phase of a weekly introduced
  practical exercise (weekly training intervention; topics: reflection on living with ease, selfcompassionate body scan, planning of positive activities, self-compassionate letter). This
  phase additionally includes smartphone reminders to apply the exercises in everyday life
  (daily training interventions).

## 2.5. SAMPLE SIZE

Previous studies from our research groups have shown a medium to large effect size for the stressor reactivity score as a primary outcome measure in online intervention studies for resilience (AG Wessa, unpublished). Because a large effect size was found only in a particularly stressed population, which is not expected in the sample addressed here, we assume a medium effect here (Hedges' g = .50). Therefore, the sample size design was calculated with a medium effect size, a significance level of 0.05 and a power of 0.90 using G\*Power (Faul et al., 2007). This results in a required sample size of n = 74 per group (N = 146). As there are high dropout rates for online interventions (van Ballegooijen et al., 2014) we decided to recruit n = 120 individuals per group. This number is based on an assumed dropout rate of 40%.

### 2.6. STUDY PROCEDURE

Once the desired sample size has been reached, a randomized controlled trial with 6 measurement time points will be conducted in which participants will be randomly assigned to either the intervention group or the waiting control group.

The intervention group receives access to the online training after randomization. The waiting control group receives access only after the first follow-up measurement (3 months after the post-measurement). Two further follow-up measurements follow (6 and 12 months after the post-measurement). The detailed time schedule can be seen in the attached flow chart. The entire data collection and intervention will be online. Neither the participants nor the study team will be blinded.



Within the practice modules, the following interventions and measurements are planned (in weeks 3 and 5, a self-care intervention is planned, in weeks 4 and 6, a self-compassion intervention is planned):

| | Practice phase: trainings and measurements (weeks 3 to 6; with buffer to complete the modules for weeks 7 & 8) | | | |
|---|---|---|---|---|
| | Day 1 | St <sub>1.1 pre</sub><br>state assessment pre-<br>intervention | Weekly intervention (approx. 30 min) | st <sub>1.1 post</sub><br>state assessment post-<br>intervention |
| | Day 2 | st <sub>1.2 pre</sub><br>state assessment pre-<br>intervention | Daily training intervention, 1st session (approx. 5-10 min) | st <sub>1.2 post</sub><br>state assessment post-<br>intervention |
| | Day 3 | st <sub>1.3 pre</sub> | Daily training intervention, 2nd session (approx. 5-10 min) | st <sub>1.3 post</sub> |
| Week 3 | Day 4 | st <sub>1.4 pre</sub> | Daily training intervention, 3rd session (approx. 5-10 min) | st <sub>1.4 post</sub> |
| | Day 5 | st <sub>1.5 pre</sub> | Daily training intervention, 4th session (approx. 5-10 min) | st <sub>1.5 post</sub> |
| | Day 6 | st <sub>1.6 pre</sub> | Daily training intervention, 5th session (approx. 5-10 min) | st <sub>1.6 post</sub> |
| | Day 7 | st <sub>1.7 pre</sub> | Daily training intervention, 6th and last session (approx. 5-10 min) | st <sub>1.7 post</sub> |
| Week 4 | Day 1 | St <sub>2.1 pre</sub><br>state assessment pre-<br>intervention | Weekly intervention (approx. 30 min) | st <sub>2.1 post</sub><br>state assessment post-<br>intervention |
| We | Day 2-7 | st <sub>2.2 pre</sub> - st <sub>2.7 pre</sub> | Daily training intervention, 2nd – 6th session (approx. 5-10 min) | st <sub>2.2 post</sub> - st <sub>2.7 post</sub> |
| Week 5 - 6 | | | | |

Legend:  $\mathsf{st}_{\mathsf{x.x\,pre}}$  = state assessment pre-intervention;  $\mathsf{st}_{\mathsf{x.x\,post}}$  = state assessment post-intervention

## 3. POPULATIONS OF ANALYSIS

We will conduct both an intention to treat (ITT) analysis as well as a per protocol (PP) analysis (see also "5.1. Statistical methodology"), with the following criteria:

## **Inclusion criteria** (included in ITT analysis):

All valid data sets

## **Exclusion criteria:**

- In PP analysis, Participants will be excluded from respective analyses if
  - they fill in less than 50% of questionnaires at a specific measurement point (e.g., pre-test) which address the primary outcome and secondary outcomes trained in the intervention
  - they fill in less than 50% of a specific questionnaire.
  - they have an implausibly short time for completing the assessments (DEG\_TIME in SoSci-Survey).
  - there is an abnormality in data (e.g., rating always the highest/ lowest on several scales).
- Participants will be excluded from the whole analysis if
  - they do not agree with the terms of usage, usage of data and privacy policy.
  - they state that their data cannot be used in a sensible way.

## 4. OUTCOME VARIABLES

## **4.1. PRIMARY OUTCOME**

• Resilience measured with *Stressor-Reactivity-Score* (SR-Score)

### 4.2. SECONDARY PARAMETERS OUTCOMES

## Outcomes related to the intervention and the primary outcome

- Resilience measured with Brief Resilience Scale (BRS; Chmitorz et al., 2018)
- Mental Health measured with General Health Questionnaire (GHQ-12; Schrnitz et al., 1999)
- Self-Compassion measured with Self-Compassion Scale Deutsch (SCS-D; Hupfeld & Ruffieux, 2011)
- Mindfulness measured with Mindful Attention and Awareness Scale (MAAS-Short; Höfling et al., 2011)
- Perceived Stress measured with Perceived Stress Scale (PSS-2+2; Schäfer et al., in preparation)
- Stressors measured with Mainz Inventory of Microstressors (MIMIS; Chmitorz et al., 2020)
- Life Events measured with Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017)
- Anxiety/ Depression measured with *Generalized Anxiety Disorder-7* (GAD-7) and *Patient Health Questionnaire*–9 (PHQ-9; Löwe et al., 2002)
- Self-Care measured with *Hamburger Selbstfürsorgefragebogen* (Hamburg Self-Care Survey; Harfst et al., 2009)
- Burnout measured with the German version of the Maslach Burnout-Inventory (MBI-D; Büssing & Perrar, 1992)
- Work-Life-Balance measured with the *Trierer Kurzskala zur Messung von Work-Life Balance* (TKS-WLB; Syrek et al., 2017)

## Further (exploratory) outcomes

- Optimism measured with Optimism-Pessimism-Scale (SOP-2; Kemper et al., 2014)
- Positive reappraisal measured with subscale of Cognitive Emotion Regulation Questionnaire (CERQ; Loch et al., 2011)
- Acceptance measured with subscale of *Cognitive Emotion Regulation Questionnaire* (CERQ; Loch et al., 2011)
- Positive (Re-)appraisal measured with Positive Appraisal Style Scale Content (PASS-content) and Positive Appraisal Style Scale Process (PASS-process; Petri-Romao et al., 2021)
- Social Support measured with Osloer Social Support Scale (OSS-3; Kocalevent et al., 2018)
- Control beliefs with Internal-External Locus of Control Short Scale—4 (IE-4; Kovaleva et al., 2014)
- Meaning measured with subscale of *Comprehensive Inventory of Thriving* (CIT; Hausler et al., 2017)

- Self-Efficacy measured with German Version of Self-Efficacy Short Scale (Allgemeine Selbstwirksamkeit Kurzskala, ASKU; Beierlein et al., 2014)
- Coping measured with *Coping Orientation to Problems Experienced Inventory* (Brief-COPE; Knoll et al., 2005)
- Self-Esteem measured with German Single-Item Self-Esteem Scale (G-SISE; Brailovskaia & Margraf, 2020)
- Positive Affect measured with subscale of Positive and Negative Affect Schedule (PANAS;
   Breyer & Bluemke, 2016)
- Life Satisfaction measured with *Satisfaction with Life Scale* (SWLS; Janke & Glöckner-Rist, 2012)
- Well-Being measured with WHO-5 Well-Being Index (Brähler et al., 2007)
- Functionality measured with World Health Organization Disability Assessment Schedule (WHODAS 2.0; Üstün et al., 2010)
- Coping Flexibility measured with Coping Flexibility Questionnaire Revised (CFQ-R; Kato, 2012)
- Satisfaction with Intervention measured with *Client Satisfaction Questionnaire-Intervention* (CSQ-I; Boß et al., 2016)
- Adverse Effects measured with *Inventory for the Assessment of Negative Effects of Psychotherapy* (INEP; Ladwig et al., 2014)
- Relationship to Intervention measured with Mobile Agnew Relationship Measure (mARM; von Wulffen et al., 2022)
- Sense of Coherence measured with Sense of Coherence Scale (SOC-29; Singer et al., 2007)
- Mental Health Literacy measured with Mental Health Literacy Questionnaire (MHLQ, Dias et al., 2018), Mental Health Literacy Scale (MHLS; O'Connor & Casey, 2015), Mental Health Knowledge Schedule (MAKS; Evans-Lacko et al., 2010), Health Literacy Survey EU 16 (HLS EU 16; Jordan & Hoebel, 2015), eHealth Literacy Scale (eHEALS; Soellner et al., 2014), Well-being Literacy Scale (Hou et al., 2021), STRESS K-10 (Giesinger et al., 2008), Fragebogen zur Erhebung des Wissens über psychosoziale Versorgungsstrukturen (Questionnaire to survey knowledge of psychosocial care structures; Fritz, 2021)
- Belief Towards Mental Illness Scale (Hirai & Clum, 2018)
- Help-seeking behaviour measured with General Help Seeking Scale (GHSS; Rickwood et al., 2005) and Attitudes Toward Seeking Professional Psychological Help (ATSPPH; Kessler et al., 2015)
- Work engagement measured with the *Utrecht Work Engagement Scale* (UWES-9; Schaufeli et al., 2006)
- Perceived work stress measured with a German translation of the Perceived Occupational Stress Scale (Marcatto et al., 2022)

#### 4.3. OTHER PARAMETERS

## **DEMOGRAPHY AND BASELINE**

## Demographic measures:

- Age
- Sex
- Educational background/ status
- Number of persons living in the household
- Number of children living in the household
- Household net income
- Individual net income

#### Baseline variables

- Attitudes towards psychological online interventions measured with Attitudes towards Psychological Online Interventions Questionnaire (APOI; Schröder et al., 2015)
- Personality measured with Big Five Inventory-10 (BFI-10; Rammstedt et al., 2017)

### Work-related variables

- Type of healthcare profession
- Number of overtime hours
- Contractually agreed working hours (full-time / part-time -> %)
- Working night shifts yes/no
- Leadership responsibility yes/no

### **USER STATISTICS**

- Intervention
- Number of processed modules (in the theory phase) and weekly and daily interventions in the practice phase
- Processing time of the individual contents as well as of the entire intervention
- Contents from the feedback questionnaire, e.g., how well the last module was liked
- Self-care, self-compassion, stress and resilience history / state queries
- Days of usage

## Survey

- Response times, namely
  - Per questionnaire (how long the user spent on each questionnaire)
  - Total processing time for all questionnaires (after adjustment for interruptions)
- Percentage of missing answers in the questionnaires (absolute and relative to total length of the survey)
- "DEG\_TIME" as normalized indicator for extremely fast completion of questionnaires

## 4.4. Hypotheses

- 1. The intervention will significantly increase resilience, measured with the SR Score, in the intervention group (IG) compared with a waitlist control (WLC) group at t₂ and t₃ compared to t₀.
- 2. The intervention will significantly increase resilience, measured with the Brief Resilience Scale, in the intervention group (IG) compared with a waitlist control (WLC) group at  $t_2$  and  $t_3$  compared to  $t_0$ .
- 3. The intervention will significantly increase self-care in the intervention group (IG) compared with a waitlist control (WLC) group at  $t_2$  and  $t_3$  compared to  $t_0$ .
- 4. The intervention will significantly increase self-compassion in the intervention group (IG) compared with a waitlist control (WLC) group at  $t_2$  and  $t_3$  compared to  $t_0$ .
- 5. The intervention will significantly increase mindfulness in the intervention group (IG) compared with a waitlist control (WLC) group at t₂ and t₃ compared to t₀.
- 6. The intervention will significantly reduce perceived stress in the intervention group (IG) compared with a waitlist control (WLC) group at  $t_2$  and  $t_3$  compared to  $t_0$
- 7. The intervention will significantly increase mental health in the intervention group (IG) compared with a waitlist control (WLC) group at  $t_2$  and  $t_3$  compared to  $t_0$ .
- 8. The intervention will significantly reduce depressive symptoms in the intervention group (IG) compared with a waitlist control (WLC) group at  $t_2$  and  $t_3$  compared to  $t_0$ .
- 9. The intervention will significantly reduce anxiety symptoms in the intervention group (IG) compared with a waitlist control (WLC) group at  $t_2$  and  $t_3$  compared to  $t_0$ .
- 10. The intervention will significantly reduce burnout symptoms in the intervention group (IG) compared with a waitlist control (WLC) group at  $t_2$  and  $t_3$  compared to  $t_0$ .
- 11. The intervention will significantly increase work-life-balance in the intervention group (IG) compared with a waitlist control (WLC) group at  $t_2$  and  $t_3$  compared to  $t_0$ .
- 12. In the intervention group, the intervention will lead to improved resilience by the end of the intervention (at  $t_2$ ) and these improvements should be maintained at the respective follow-ups (at  $t_3$ ,  $t_4$ ,  $t_5$ ; probably to a lesser degree).
- 13. Self-compassion interventions (weekly intervention and daily training intervention) in the practice modules:
  - A) For the weekly interventions, the state self-compassion measure will be significantly higher after the interventions (comparison of  $st_{2.1pre}$  vs.  $st_{2.1post}$  and  $st_{4.1pre}$  vs.  $st_{4.1post}$ ).
  - B) For the first session of the daily training interventions, the state self-compassion measure will be significantly higher after the interventions (comparison of st<sub>2.2pre</sub> vs. st<sub>2.2post</sub> and st<sub>4.2pre</sub> vs. st<sub>4.2post</sub>).
- 14. Self-care interventions (weekly intervention and daily training intervention) in the practice modules:
  - A) For the weekly interventions, the state self-compassion measure will be significantly higher after the interventions (comparison of  $st_{1.1pre}$  vs.  $St_{1.1post}$  and  $st_{3.1pre}$  vs.  $st_{3.1post}$ ).
  - B) For the first session of the daily training interventions, the state self-compassion measure will be significantly higher after the interventions (comparison of  $st_{1.2pre}$  vs.  $st_{1.2post}$  and  $st_{3.2pre}$  vs.  $st_{3.2post}$ ).
- 15. For the intervention group, the number of weekly interventions and daily training interventions completed will result in a significant
  - A) increase of self-care at t2
  - B) increase of self-compassion at t<sub>2</sub>
  - C) increase of resilience measured with SR score at t<sub>2</sub>
  - D) decrease of burnout symptoms at t<sub>2</sub>

Further longitudinal effects, intervention effects at intermediate measurements ( $t_1$ ), other resilience-related outcomes as well as moderator and mediator analyses will be examined exploratorily. Therefore, no specific hypotheses are stated.

## 5. STATISTICAL METHODOLOGY

#### **5.1. GENERAL METHODOLOGY**

Demographics and work-related variables will be reported with means and standard deviations for continuous variables (e.g., age) and as frequencies for categorial variables (e.g., gender). Items of questionnaires (e.g., Sense of Coherence Scale) will be recoded (where applicable) and a scale mean or sum score will be calculated in data processing. Means/sum scores and standard deviations will be reported separately by treatment group. If applicable, means and standard deviations of user statistics will be calculated and reported (e.g., means among the subgroup of users who completed a specific module). For continuous outcomes, we will use t-tests for independent samples and for categorical outcome we will employ  $\chi^2$ -tests to examine baseline differences between training and control

#### HANDLING OF MISSING DATA

group in demographic data or measured variables.

- On the one hand, the data will be analysed according to the "intention-to-treat" principle, with missing values being replaced using appropriate imputation methods.
- On the other hand, the results will be reported as "per-protocol" analysis, in which only those cases are considered that have gone through the study procedure as defined by protocol. We consider the intervention to be completed for participants who, in addition to the theory modules, completed at least 50% of the weekly interventions and the daily training interventions. To note, a maximum of 4 weekly interventions with 6 daily interventions can be reached. In the per-protocol analysis, only these participants will be included. To control for influences of compliance, usage of intervention will be examined as covariate in an exploratory analysis.

## **CLASSIFICATION OF PROTOCOL VIOLATION**

Exclusion of participants due to protocol violations will be reported in the methods / results section. To examine outliers in the questionnaire data, boxplots will be created.

## **5.2. PRIMARY AND SECONDARY DATA ANALYSES**

In primary and secondary data analyses, all stated hypotheses will be tested. In all analyses an error probability of  $\alpha$  = .05 will be set a priori for interference statistics calculations. In cases of multiple testing,  $\alpha$  will be adjusted accordingly. In addition to statistical significance, descriptive statistics and effect sizes (e.g., Cohen's d) will be reported. Publication of results will follow CONSORT guidelines for transparent reporting of randomized trials.

Cronbach's  $\alpha$  and McDonald's  $\omega$  will be calculated as measure of reliability of the respective questionnaires.

Before data analysis, assumptions of statistical methods (e.g., variance of homogeneity, normal distribution) will be tested with suitable procedures (e.g., Levene-tests, Box's M, histograms, QQ-plots, and Shapiro-Wilk-Test). Zero-order correlations between study variables will be reported. Non-parametric correlation calculation will be based on results of (non-)normality, etc. Variables will be standardized where applicable.

The analysis plan for H1 to H11 is as follows:

- Differences between study groups in primary and secondary outcomes before (t<sub>0</sub>) and after the intervention (t<sub>2</sub>) and at the time of the first follow-up (t<sub>3</sub>) will be examined using mixed analyses of covariance (ANCOVA), with group (intervention vs. waitlist-control) as a between-subjects factor, time (t<sub>0</sub>, t<sub>2</sub>, t<sub>3</sub>) as a within-subjects factor and pre-measurement (t<sub>0</sub>) included as a covariate to increase test power. Outcomes will be the primary outcome resilience (measured with SR Score) and the secondary outcomes resilience (measured with BRS), perceived stress, self-care, self-compassion, mindfulness, mental health, depression, anxiety, burnout, and work-life-balance, respectively.
- If applicable, post-hoc *t*-tests will be conducted.
- Effect sizes will be calculated for the ANCOVA (i.e., Eta<sup>2</sup>) as well as for between-group differences (i.e., Cohen's d) at post-intervention assessment (t<sub>2</sub>) and the first follow-up assessment (t<sub>3</sub>). Also, the effect size of the intervention effect will be calculated (i.e., Cohen's d).

The analysis plan for H12 is as follows: term effect over the follow-up measurements ( $t_0$  to  $t_5$ ) within the intervention group will be tested using a repeated measures ANOVA.

- If applicable, post-hoc *t*-tests and planned contrasts will be conducted.
- Effect sizes will be calculated.
- Eta<sup>2</sup> will be calculated as measure for effect size for the ANOVA.

The analysis plan for H13 and H14 is as follows:

- In order to test whether the changes in the state measurements (pre- to post-intervention in state self-compassion and state self-care) are significant, we will conduct within-group *t*-tests. We will perform separate tests for state self-compassion and state self-care, each for (1) the weekly training interventions and (2) the first practice of daily interventions, respectively.
- Cohen's d will be calculated as measure for effect size.

The analysis plan for H15 is as follows:

- Linear regressions will be conducted with the following predictor and criterion variables:
  - Predictor variables:
    - baseline-values of self-care (and, in separate models, self-compassion / resilience / burnout, respectively) at t<sub>0</sub>
    - amount of interventions completed (number of weekly training interventions and daily interventions)

- Criterion variables:
  - Post-intervention values of self-care (and, in separate models, self-compassion / resilience / burnout, respectively) at t<sub>2</sub>

If assumptions for the mentioned statistical methods are violated, appropriate non-parameteric statistical methods will be chosen.

### **5.3. EXPLORATORY DATA ANALYSES**

All other outcome measures mentioned above and not directly addressed in the intervention will be evaluated exploratively.

In addition, changes will be examined in correlative network analyses of the variables. Moderator and mediator analyses are intended as exploratory analyses to examine the influence of mediating/moderating variables (e.g., gender, personality, intervention usage, attitudes toward online psychological interventions, coping styles) of the primary correlations.

The intermediate survey  $(t_1)$  will be exploratively included in the analyses.

#### References

- Beierlein, C., Kovaleva, A., Kemper, C. J., & Rammstedt, B. (2014). Allgemeine Selbstwirksamkeit Kurzskala (ASKU). *Zusammenstellung sozialwissenschaftlicher Items und Skalen (ZIS)*. https://doi.org/10.6102/ZIS35
- Boß, L., Lehr, D., Reis, D., Vis, C., Riper, H., Berking, M., & Ebert, D. D. (2016). Reliability and Validity of Assessing User Satisfaction With Web-Based Health Interventions. *Journal of Medical Internet Research*, *18*(8), e234. https://doi.org/10.2196/jmir.5952
- Brähler, E., Mühlan, H., Albani, C., & Schmidt, S. (2007). Teststatistische Prüfung und Normierung der deutschen Versionen des EUROHIS-QOL Lebensqualität-Index und des WHO-5 Wohlbefindens-Index. *Diagnostica*, *53*(2), 83–96. https://doi.org/10.1026/0012-1924.53.2.83
- Brailovskaia, J., & Margraf, J. (2020). How to measure self-esteem with one item? Validation of the German single-item self-esteem scale (G-SISE). *Current Psychology*, *39*(6), 2192–2202. https://doi.org/10.1007/s12144-018-9911-x
- Breyer, B., & Bluemke, M. (2016). Deutsche Version der Positive and Negative Affect Schedule PANAS (GESIS Panel). *Zusammenstellung sozialwissenschaftlicher Items und Skalen (ZIS*). https://doi.org/10.6102/ZIS242
- Büssing, A., & Perrar, K. M. (1992). Die Messung von Burnout. Untersuchung einer deutschen Fassung des Malach Burnout Inventars. *Diagnostica*, *38*(4), 328–353.
- Chmitorz, A., Kurth, K., Mey, L. K., Wenzel, M., Lieb, K., Tüscher, O., Kubiak, T., & Kalisch, R. (2020).

  Assessment of Microstressors in Adults: Questionnaire Development and Ecological Validation of the Mainz Inventory of Microstressors. *JMIR Mental Health*, 7(2), e14566.

  https://doi.org/10.2196/14566
- Chmitorz, A., Wenzel, M., Stieglitz, R.-D., Kunzler, A., Bagusat, C., Helmreich, I., Gerlicher, A., Kampa, M., Kubiak, T., Kalisch, R., Lieb, K., & Tüscher, O. (2018). Population-based validation of a German version of the Brief Resilience Scale. *PLOS ONE*, *13*(2), e0192761. https://doi.org/10.1371/journal.pone.0192761

- Corrigan, P. W., Michaels, P. J., Vega, E., Gause, M., Watson, A. C., & Rüsch, N. (2012). Self-stigma of mental illness scale—short form: Reliability and validity. *Psychiatry Research*, *199*(1), 65–69. https://doi.org/10.1016/j.psychres.2012.04.009
- Dias, P., Campos, L., Almeida, H., & Palha, F. (2018). Mental Health Literacy in Young Adults: Adaptation and Psychometric Properties of the Mental Health Literacy Questionnaire. *International Journal of Environmental Research and Public Health*, *15*(7), 1318. https://doi.org/10.3390/ijerph15071318
- Evans-Lacko, S., Little, K., Meltzer, H., Rose, D., Rhydderch, D., Henderson, C., & Thornicroft, G. (2010).

  Development and Psychometric Properties of the Mental Health Knowledge Schedule. *The*Canadian Journal of Psychiatry, 55(7), 440–448. https://doi.org/10.1177/070674371005500707
- Faul, F., Erdfelder, E., Lang, A.-G., & Buchner, A. (2007). G\*Power 3: A flexible statistical power analysis program for the social, behavioral, and biomedical sciences. *Behavior Research Methods*, *39*(2), 175–191. https://doi.org/10.3758/BF03193146
- Fritz, B. (2021). Seelsorge mit psychisch kranken Menschen und Vernetzung der Seelsorgenden mit der psychosozialen Gesundheitsversorgung der BRD [Bachelorarbeit]. Philipps-Universität Marburg.
- Giesinger, J., Rumpold, Mag. G., & Schüßler, G. (2008). Die K10-Screening-Skala für unspezifischen psychischen Distress. *Psychosomatik und Konsiliarpsychiatrie*, *2*(2), 104–111. https://doi.org/10.1007/s11800-008-0100-x
- Hausler, M., Huber, A., Strecker, C., Brenner, M., Höge, T., & Höfer, S. (2017). Validierung eines

  Fragebogens zur umfassenden Operationalisierung von Wohlbefinden: Die deutsche Version des

  Comprehensive Inventory of Thriving (CIT) und die Kurzversion Brief Inventory of Thriving (BIT).

  Diagnostica, 63(3), 219–228. https://doi.org/10.1026/0012-1924/a000174
- Höfling, V., Moosbrugger, H., Schermelleh-Engel, K., & Heidenreich, T. (2011). Mindfulness or Mindlessness?: A Modified Version of the Mindful Attention and Awareness Scale (MAAS). *European Journal of Psychological Assessment*, 27(1), 59–64. https://doi.org/10.1027/1015-5759/a000045

- Hou, H., Chin, T.-C., Slemp, G. R., & Oades, L. G. (2021). Wellbeing Literacy: Conceptualization,
  Measurement, and Preliminary Empirical Findings from Students, Parents and School Staff.
  International Journal of Environmental Research and Public Health, 18(4), 1485.
  https://doi.org/10.3390/ijerph18041485
- Hupfeld, J., & Ruffieux, N. (2011). Validierung einer deutschen Version der Self-Compassion Scale (SCS-D).

  Zeitschrift für Klinische Psychologie und Psychotherapie, 40(2), 115–123.

  https://doi.org/10.1026/1616-3443/a000088
- Janke, S., & Glöckner-Rist, A. (2012). Deutsche Version der Satisfaction with Life Scale (SWLS).

  Zusammenstellung sozialwissenschaftlicher Items und Skalen (ZIS). https://doi.org/10.6102/ZIS147
- Jordan, S., & Hoebel, J. (2015). Gesundheitskompetenz von Erwachsenen in Deutschland: Ergebnisse der Studie "Gesundheit in Deutschland aktuell" (GEDA). *Bundesgesundheitsblatt Gesundheitsforschung Gesundheitsschutz, 58*(9), 942–950. https://doi.org/10.1007/s00103-015-2200-z
- Kato, T. (2012). Development of the Coping Flexibility Scale: Evidence for the coping flexibility hypothesis.

  \*\*Journal of Counseling Psychology, 59(2), 262–273. https://doi.org/10.1037/a0027770
- Kemper, C. J., Beierlein, C., Kovaleva, A., & Rammstedt, B. (2014). *Eine Kurzskala zur Messung von Optimismus-Pessimismus*. GESIS Leibniz-Institut für Sozialwissenschaften.
- Kessler, E.-M., Agines, S., & Bowen, C. E. (2015). Attitudes towards seeking mental health services among older adults: Personal and contextual correlates. *Aging & Mental Health*, *19*(2), 182–191. https://doi.org/10.1080/13607863.2014.920300
- Knoll, N., Rieckmann, N., & Schwarzer, R. (2005). Coping as a mediator between personality and stress outcomes: A longitudinal study with cataract surgery patients. *European Journal of Personality*, 19(3), 229–247. https://doi.org/10.1002/per.546

- Kocalevent, R.-D., Berg, L., Beutel, M. E., Hinz, A., Zenger, M., Härter, M., Nater, U., & Brähler, E. (2018).

  Social support in the general population: Standardization of the Oslo social support scale (OSSS-3).

  BMC Psychology, 6(1), 31. https://doi.org/10.1186/s40359-018-0249-9
- Kovaleva, A., Beierlein, C., Kemper, C. J., & Rammstedt, B. (2014). Internale-Externale-Kontrollüberzeugung-4 (IE-4). Zusammenstellung sozialwissenschaftlicher Items und Skalen (ZIS).

  https://doi.org/10.6102/ZIS184
- Krüger-Gottschalk, A., Knaevelsrud, C., Rau, H., Dyer, A., Schäfer, I., Schellong, J., & Ehring, T. (2017). The German version of the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Psychometric properties and diagnostic utility. *BMC Psychiatry*, *17*(1), 379. https://doi.org/10.1186/s12888-017-1541-6
- Ladwig, I., Rief, W., & Nestoriuc, Y. (2014). Welche Risiken und Nebenwirkungen hat Psychotherapie? Entwicklung des Inventars zur Erfassung Negativer Effekte von Psychotherapie (INEP).

  Verhaltenstherapie, 24(4), 252–263. https://doi.org/10.1159/000367928
- Loch, N., Hiller, W., & Witthöft, M. (2011). Der Cognitive Emotion Regulation Questionnaire (CERQ): Erste teststatistische Überprüfung einer deutschen Adaption. *Zeitschrift für Klinische Psychologie und Psychotherapie*, *40*(2), 94–106. https://doi.org/10.1026/1616-3443/a000079
- Löwe, B., Spitzer, R. L., Zipfel, S., & Herzog, W. (2002). *Gesundheitsfragebogen für Patienten (PHQ-D). Manual und Testunterlagen.* (2. Auflage). Pfizer.
- Marcatto, F., Di Blas, L., Luis, O., Festa, S., & Ferrante, D. (2022). The Perceived Occupational Stress Scale: A

  Brief Tool for Measuring Workers' Perceptions of Stress at Work. *European Journal of Psychological*Assessment, 38(4), 293–306. https://doi.org/10.1027/1015-5759/a000677
- O'Connor, M., & Casey, L. (2015). The Mental Health Literacy Scale (MHLS): A new scale-based measure of mental health literacy. *Psychiatry Research*, *229*(1–2), 511–516.

  https://doi.org/10.1016/j.psychres.2015.05.064

- Petri-Romao, P., Ropanova, A., Tuescher, O., Basten, U., & Kalisch, R. (2021, September 29). *Positive*Appraisal Style Scales—Development and validation of self-report assessment of positive appraisal style. Resilience Symposium 2021, Mainz.
- Rammstedt, B., Kemper, C. J., Klein, M. C., Beierlein, C., & Kovaleva, A. (2017). A Short Scale for Assessing the Big Five Dimensions of Personality: 10 Item Big Five Inventory (BFI-10). *Methoden, Daten, Analysen*, 7(2), 233–249. https://doi.org/10.12758/MDA.2013.013
- Rickwood, D., Deane, F. P., Wilson, C. J., & Ciarrochi, J. (2005). Young people's help-seeking for mental health problems. *Australian E-Journal for the Advancement of Mental Health*, *4*(3), 218–251. https://doi.org/10.5172/jamh.4.3.218
- Schäfer, S. K., von Boros, L., Göritz, A. S., Baumann, S., Tüscher, O., Lieb, K., & Möhring. (in preparation). *The Perceived Stress Scale 2&2: A Two-Factorial German Short Version of the Perceived Stress Scale*.
- Schaufeli, W. B., Bakker, A. B., & Salanova, M. (2006). The Measurement of Work Engagement With a Short

  Questionnaire: A Cross-National Study. *Educational and Psychological Measurement*, *66*(4), 701–716. https://doi.org/10.1177/0013164405282471
- Schrnitz, N., Kruse, J., & Tress, W. (1999). Psychometric properties of the General Health Questionnaire (GHQ-12) in a German primary care sample. *Acta Psychiatrica Scandinavica*, 100(6), 462–468. https://doi.org/10.1111/j.1600-0447.1999.tb10898.x
- Schröder, J., Sautier, L., Kriston, L., Berger, T., Meyer, B., Späth, C., Köther, U., Nestoriuc, Y., Klein, J. P., & Moritz, S. (2015). Development of a questionnaire measuring Attitudes towards Psychological Online Interventions—the APOI. *Journal of Affective Disorders*, *187*, 136—141. https://doi.org/10.1016/j.jad.2015.08.044
- Singer, S., Brähler, E., & Schumacher, J. (2007). *Die "Sense of Coherence Scale": Testhandbuch zur deutschen Version*. Vandenhoeck & Ruprecht.

- Soellner, R., Huber, S., & Reder, M. (2014). The Concept of eHealth Literacy and Its Measurement: German

  Translation of the eHEALS. *Journal of Media Psychology*, 26(1), 29–38.

  https://doi.org/10.1027/1864-1105/a000104
- Syrek, C. J., Weigelt, O., Peifer, C., & Antoni, C. H. (2017). Zeigarnik's sleepless nights: How unfinished tasks at the end of the week impair employee sleep on the weekend through rumination. *Journal of Occupational Health Psychology*, 22(2), 225–238. https://doi.org/10.1037/ocp0000031
- Üstün, T. B., Chatterji, S., Kostanjsek, N., Rehm, J., Kennedy, C., Epping-Jordan, J., Saxena, S., von Korff, M., & Pull, C. (2010). Developing the World Health Organization Disability Assessment Schedule 2.0.

  \*\*Bulletin of the World Health Organization, 88(11), 815–823. https://doi.org/10.2471/BLT.09.067231
- van Ballegooijen, W., Cuijpers, P., van Straten, A., Karyotaki, E., Andersson, G., Smit, J. H., & Riper, H.

  (2014). Adherence to Internet-Based and Face-to-Face Cognitive Behavioural Therapy for

  Depression: A Meta-Analysis. *PLoS ONE*, *9*(7), e100674.

  https://doi.org/10.1371/journal.pone.0100674
- von Wulffen, C., Marciniak, M. A., Rohde, J., Kalisch, R., Binder, H., Tüscher, O., & Kleim, B. (2022). *German version of the mobile Agnew Relationship Measure (mARM-G): Translation and validation study*[Preprint]. PsyArXiv. https://doi.org/10.31234/osf.io/76gey